CLINICAL TRIAL: NCT03526341
Title: Post Market Clinical Follow Up Study for ReliaTack™ Articulating Reloadable Fixation Device With Deep Purchase Tacks
Acronym: RAFDT
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17047RAF
Record Dates: First submitted 2018-04-17; First posted 2018-05-16 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Inguinal Hernia; Ventral Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: ReliaTack™ Articulating Reloadable Fixation Device — ReliaTack™ Articulating Reloadable Fixation Device with Deep Purchase Tacks

SUMMARY:
A post-market clinical follow-up study for ReliaTack™ articulating reloadable fixation device with deep purchase tacks

DETAILED DESCRIPTION:
A retrospective, multi-center, chart review of medical records on the use of the device for two (2) surgical procedure indications:

1. inguinal/femoral hernia
2. ventral hernia

A minimum of 4 sites in the United States will perform chart review and enter 116 study records in the database for data collection. The 116 subject records will be comprised of 76 for the inguinal/femoral indication, and 40 for the ventral indication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject underwent ventral or inguinal/femoral hernia repair procedure utilizing ReliaTack™ Articulating Reloadable Fixation Device with Deep Purchase Tacks on or after 510(k) approval.
2. Medical records are available, which document a ventral and/or inguinal/femoral hernia repair surgical procedure.

Exclusion Criteria:

1. Institutional Review Board (IRB) consent requirement cannot be met:

   1. waiver of subject informed consent requirements are not granted by IRB* and,
   2. an altercation to the consent process is not granted by the IRB and,
   3. subject or subject's parent or legal guardian is unable or unwilling to provide signed informed consent
2. Subject was participating in any investigational drug or device study at the time of surgery or within 30-day (+3 days) study window
3. Subject was pregnant at the time of procedure
4. Subject had a documented allergy at the time of surgery to any of the components of the device or the mesh implant
5. Subject was treated with any other implantable mechanical fixation device, other than sutures

   * A waiver of subject informed consent procedures will be requested from all IRBs of record for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who previously underwent minimally invasive or open surgical ventral or inguinal/femoral hernia repair procedures using the ReliaTack™ Articulating Reloadable Fixation Device with Deep Purchase Tacks.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
To confirm the safety for this device during inguinal/ femoral and ventral hernia repair procedures by assessing the proportion of subjects with SADE's/AEs | 30 days (+3 days) post procedure
  Safety will be assessed as the proportion of subjects with SADE's/AEs

SECONDARY OUTCOMES:
The rate of device-related malfunctions will be captured to confirm the performance for this device during inguinal/ femoral and ventral hernia repair procedures | 30 days (+3 days) post procedure
  The rate of device-related malfunctions affecting performance of the device will be captured

CONTACTS AND LOCATIONS:
Overall Officials: John W Odom, MD, Principal Investigator — St. Josephs/ Candler; Har Chi Lau, MD, Principal Investigator — Hudson Valley Surgical Group
Locations (1):
- Hudson Valley Surgical Group, Sleepy Hollow, New York, United States

IPD SHARING:
Plan to Share IPD: No